CLINICAL TRIAL: NCT05755100
Title: I MOVE!+UP: Piloting an Integrated Weight Management Program for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Hoerster, Principal Investigator, VA Puget Sound Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1670114
Record Dates: First submitted 2023-02-08; First posted 2023-03-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: PTSD; Overweight and Obesity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Uncontrolled pilot trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot study of I MOVE!+UP among Veterans with PTSD and BMI of 30 or greater. (Other): Single arm pilot trial.
  Interventions: Behavioral: I MOVE!+UP

INTERVENTIONS:
Behavioral: I MOVE!+UP — An individual psychotherapy that integrates behavioral weight management with evidence-based psychotherapy for PTSD (Cognitive Processing Therapy) for up to 6 months, augmented with evidence-based psychiatric and weight management medication management.

SUMMARY:
This study seeks to test I MOVE!+UP, which integrates individual evidence-based psychotherapy for PTSD with behavioral weight management among Veterans with a Body Mass Index of at least 30 and meeting criteria for current PTSD. Participants will continue receiving routine primary care and psychiatric care management as indicated, in coordination with the I MOVE!+UP therapist. This study is being conducted to see whether I MOVE!+UP holds promise as a treatment for commonly co-occurring PTSD and high Body Mass Index. Participation will involve attending up to 16 psychotherapy visits that last approximately 1-2 hours over 6 months and attending 2 study assessment visits that last approximately 1-2 hours at enrollment and 6 months. Active participation will take up to approximately 6 months.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD), prevalent among Veterans, puts Veterans at increased risk for obesity and related conditions. Veterans with PTSD lose less weight in VA's MOVE! weight management program, due to PTSD symptoms that interfere with activity and healthy diet. In addition, many Veterans who receive evidence-based PTSD treatment remain symptomatic. A behavioral weight loss program that augments standard PTSD care and targets PTSD-related weight loss barriers called MOVE!+UP was piloted and iteratively refined among 44 overweight Veterans with PTSD, and is currently being tested in an RCT. However, not all Veterans will participate in group-based treatment and prior work on integrated tobacco cessation with individual psychotherapy was quite impactful, and was particularly well-suited for coordinating augmentative medication management using shared decision-making. As such, we propose to conduct an uncontrolled pilot of an intervention called I MOVE!+UP. It will integrate MOVE!+UP into individual evidence-based psychotherapy (i.e.., Cognitive Processing Therapy) for PTSD for up to 6 months, augmented with evidence-based psychiatric and weight management medication management coordination. If I MOVE!+UP is acceptable, feasible, and proof-of-concept outcomes demonstrate potential benefit to weight and PTSD outcomes, we will apply for large-scale funding to test it in an RCT. I MOVE!+UP integrated behavioral intervention will be led by a psychotherapist (social worker, psychologist, or trainee in those disciplines). Because this care will be delivered within the context of routine mental health care, patients will be offered the opportunity for individualized pharmacotherapy for weight loss and psychiatric symptom management as part of their care plan.

ELIGIBILITY:
Inclusion Criteria:

* - U.S. military Veteran

  * PTSD Diagnosis: standard criteria for PTSD Checklist for DSM-5 (PCL-5): lifetime.
* - Experience of trauma, a score of ≥33, and meets criteria for the symptom domains.
* - Body Mass Index (BMI) of ≥ 30 kg/m2.
* - Willing to participate in all intervention and assessment activities

Exclusion Criteria:

* - Not fluent in English, severe hearing loss, no phone access.
* - Current MOVE! participation (at least 2 sessions in the past 3 months.)
* - Current PTSD psychotherapy participation (at least 2 PE or CPT sessions in the past 3 months.)
* - Past year bariatric surgery or planning to have bariatric surgery in next 6 months.
* - Current pregnancy.
* - Based on clinical judgment, would be unable to participate because of a) acutely exacerbated substance use, mental health, or chronic medical conditions or b) moderate to severe chronic, progressive neurologic conditions such as Dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Weight | change from baseline to 6 months
  in person weight taken during research visit
PTSD symptoms | change from baseline to 6 months
  PCL-5 (self-reported)

SECONDARY OUTCOMES:
Depression symptoms | change from baseline to 6 months
  PhQ-8 (self-reported)
Insomnia severity | change from baseline to 6 months
  Insomnia severity index (self-reported)
Diet quality | change from baseline to 6 months
  Starting the Conversation (self-reported)
Social support for physical activity and healthy eating | change from baseline to 6 months
  Modified based on Sallis et al measure (self-reported)
Internalized weight bias | change from baseline to 6 months
  Internalized weight bias measure (self-reported)
Health-related quality of life | change from baseline to 6 months
  Sf-12 (self-reported)
Waist circumference | change from baseline to 6 months
  In person, taken during research visit
Blood pressure (systolic) | change from baseline to 6 months
  In person, taken during research visit
Blood pressure (diastolic) | change from baseline to 6 months
  In person, taken during research visit
Total cholesterol | change from baseline to 6 months
  In person, bloodwork taken during research visit
LDL cholesterol | change from baseline to 6 months
  In person, bloodwork taken during research visit
HDL cholesterol | change from baseline to 6 months
  In person, bloodwork taken during research visit
Triglycerides | change from baseline to 6 months
  In person, bloodwork taken during research visit
HbA1C | change from baseline to 6 months
  In person, bloodwork taken during research visit

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Hoerster, PhD, MPH, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States